CLINICAL TRIAL: NCT00051051
Title: A Phase II, Randomized, Open-Label Study of Single Agent CI-1033 in Patients With Metastatic Breast Cancer
Brief Title: A Phase II Study of CI-1033 in Treating Patients With Metastatic (Stage IV) Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1033-011
Record Dates: First submitted 2003-01-02; First posted 2003-01-03 (Estimated); Last update posted 2007-05-04 (Estimated); Status verified 2006-09

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Canertinib

INTERVENTIONS:
Drug: CI-1033

SUMMARY:
CI-1033 is an experimental drug that acts as an inhibitor of erbB (EGFR) receptors, which may be involved in tumor growth. The primary objective of this study is to assess the antitumor activity of CI-1033 in patients with metastatic breast cancer. Patients with histologically confirmed metastatic (Stage IV) breast cancer and who have received no more than 2 prior cytotoxic chemotherapy regimens are eligible for this study. CI-1033 is administered orally. Patients are required to have blood tests periodically while receiving treatment and will be closely monitored throughout the study for possible side effects and response to treatment. Patients may not have received any prior treatment with other agents that target erbB receptors, including Herceptin (trastuzumab) or Iressa (gefitinib).

ELIGIBILITY:
Inclusion Criteria:

* Female, at least 18 years of age
* Histologically confirmed diagnosis of breast cancer
* Metastatic (Stage IV) disease
* Progressive or recurrent disease following the most recent therapy
* No more than 2 different, prior cytotoxic chemotherapy regimens for metastatic disease
* At least one measurable target lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) that has not been irradiated
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, determined within 2 weeks prior to randomization
* Estimated life expectancy of > 12 weeks
* Capable of giving written informed consent
* Capable of swallowing intact CI-1033 capsules
* Capable of understanding and adhering to the protocol requirements
* No prior exposure to CI-1033 or other agents that target the erbB receptor family (such as Herceptin, Iressa, Tarceva, IMC-C225, and EKB-569)
* No known hypersensitivity reaction to tyrosine kinase inhibitors
* Adequate liver, renal, or bone marrow function determined within 2 weeks prior to randomization
* No cytotoxic chemotherapy within 3 weeks prior to baseline disease assessments (6 weeks for nitrosoureas or mitomycin)
* No immunotherapy (including Herceptin) or other biologic therapy within 2 weeks prior to baseline disease assessments
* No hormone therapy (including hormone replacement therapy) within 4 weeks prior to baseline disease assessments (6 weeks for megestrol acetate)
* Patients must have recovered from the acute effects of any radiation therapy or surgery
* No treatment with any other investigational therapy within 4 weeks prior to baseline disease assessments
* No history of any cancer other than the present condition (except nonmelanoma skin cancer or carcinoma in situ of the cervix) within the last 5 years
* No patients with untreated brain metastases or patients that have not recovered from treatment for brain metastases
* No known malabsorption syndrome or other condition that may impair absorption of study medication
* No comorbidity or condition which compromises compliance with this protocol as judged by the investigator or that would significantly complicate interpretation of the safety profile of CI-1033
* No patients having reproductive potential who are not using a method of birth control or who are pregnant or breastfeeding or have a positive pregnancy test during baseline

Exclusion Criteria:

Prior exposure to CI-1033 or other agents that target the erbB receptor family; cytotoxic chemotherapy within 3 weeks prior to baseline disease assessments (6 weeks for nitrosoureas or mitomycin); immunotherapy (including Herceptin) or other biologic therapy within 2 weeks prior to baseline disease assessments; hormone therapy (including hormone replacement therapy) within 4 weeks prior to baseline disease assessments; 6 weeks for megestrol acetate (to exclude the possibility of a hormone-withdrawal response); patients with untreated brain metastases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168
Dates: Start 2002-12; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
The primary objective is to assess the antitumor activity of CI 1033 in patients with metastatic breast cancer.

SECONDARY OUTCOMES:
Secondary objectives include an assessment of safety and patient reported outcomes (eg, quality of life [QOL])
correlations between erbB expression and efficacy
exploratory analyses of soluble erbB-2 or other biomarkers
exploratory questions to measure the patient-reported impact of diarrhea and skin reactions will also be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (53):
- United States (34):
  - Pfizer Investigational Site, Montgomery, Alabama
  - Pfizer Investigational Site, Arroyo Grande, California
  - Pfizer Investigational Site, Montebello, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Aventura, Florida
  - Pfizer Investigational Site, Miami Beach, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Maywood, Illinois
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Lenexa, Kansas
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Brownstown, Michigan
  - Pfizer Investigational Site, Dearborn, Michigan
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, West Bloomfield, Michigan
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Lee's Summit, Missouri
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Gallatin, Tennessee
  - Pfizer Investigational Site, Hermitage, Tennessee
  - Pfizer Investigational Site, Lebanon, Tennessee
  - Pfizer Investigational Site, Murfreesboro, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Walla Walla, Washington
- Belgium (2):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Leuven
- Canada (4):
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Chicoutimi, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
- France (2):
  - Pfizer Investigational Site, Avignon
  - Pfizer Investigational Site, Paris
- Ireland (2):
  - Pfizer Investigational Site, Dublin
  - Pfizer Investigational Site, Galway
- Italy (4):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Forlì
  - Pfizer Investigational Site, Modena
  - Pfizer Investigational Site, Roma
- Pfizer Investigational Site, Madrid, Madrid, Spain
- Pfizer Investigational Site, Stockholm, Sweden
- United Kingdom (3):
  - Pfizer Investigational Site, Sutton, Surrey
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, London

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=1033-011&StudyName=A+Phase+II+Study+of+CI%2D1033+in+Treating+Patients+with+Metastatic+%28Stage+IV%29+Breast+Cancer